CLINICAL TRIAL: NCT00569634
Title: Agreement Between Venous and Arterial Blood Gas Measurements in the Intensive Care Unit
Acronym: AVANTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07H-821001
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Acid-Base Balance
Keywords: Venous blood gas; Arterial blood gas; pH; pCO2; Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Venous blood gas analysis

INTERVENTIONS:
Procedure: Venous blood gas analysis — When an ABG is deemed to be necessary as part of ICU management, a central venous sample will also be obtained with minimum delay (always < 2 minutes) between the samples. The samples will be analyzed by a blood gas analyzer as quickly as possible.

SUMMARY:
The purpose of this study is to examine the agreement between venous blood gas and arterial blood gas measurements in patients in the Intensive Care Unit.

DETAILED DESCRIPTION:
Venous blood gas analysis may be an alternative to arterial blood gas analysis for acid-base status, reducing the need for frequent invasive arterial sampling. The objective of this study is to examine the agreement between ABG and VBG samples for all commonly used parameters (pH, pCO2 and bicarbonate) in a pathologically diverse ICU patient population, specifically analyzing multiple paired arterial and venous samples from each patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years or older
* Admitted to the Intensive Care Unit (ICU)
* Determined by their treating clinicians to require both a central venous line and arterial line

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Agreement between venous and arterial blood gas measurements of pH, pCO2 and bicarbonate | Duration of Intensive Care Unit Admission

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Treger, M.D., Principal Investigator — Olive View-UCLA Education & Research Institute

REFERENCES:
- [Background] Mortensen JD. Clinical sequelae from arterial needle puncture, cannulation, and incision. Circulation. 1967 Jun;35(6):1118-23. doi: 10.1161/01.cir.35.6.1118. No abstract available. PMID 6026202
- [Background] Criscuolo C, Nepper G, Buchalter S. Reflex sympathetic dystrophy following arterial blood gas sampling in the intensive care setting. Chest. 1995 Aug;108(2):578-80. doi: 10.1378/chest.108.2.578. PMID 7634906
- [Background] Malinoski DJ, Todd SR, Slone S, Mullins RJ, Schreiber MA. Correlation of central venous and arterial blood gas measurements in mechanically ventilated trauma patients. Arch Surg. 2005 Nov;140(11):1122-5. doi: 10.1001/archsurg.140.11.1122. PMID 16342377
- [Background] Kelly AM, Kyle E, McAlpine R. Venous pCO(2) and pH can be used to screen for significant hypercarbia in emergency patients with acute respiratory disease. J Emerg Med. 2002 Jan;22(1):15-9. doi: 10.1016/s0736-4679(01)00431-0. PMID 11809551
- [Background] Rang LC, Murray HE, Wells GA, Macgougan CK. Can peripheral venous blood gases replace arterial blood gases in emergency department patients? CJEM. 2002 Jan;4(1):7-15. doi: 10.1017/s1481803500006011. PMID 17637143
- [Background] Kelly AM, McAlpine R, Kyle E. Agreement between bicarbonate measured on arterial and venous blood gases. Emerg Med Australas. 2004 Oct-Dec;16(5-6):407-9. doi: 10.1111/j.1742-6723.2004.00642.x. PMID 15537402
- [Background] Kelly AM, McAlpine R, Kyle E. Venous pH can safely replace arterial pH in the initial evaluation of patients in the emergency department. Emerg Med J. 2001 Sep;18(5):340-2. doi: 10.1136/emj.18.5.340. PMID 11559602
- [Background] Ma OJ, Rush MD, Godfrey MM, Gaddis G. Arterial blood gas results rarely influence emergency physician management of patients with suspected diabetic ketoacidosis. Acad Emerg Med. 2003 Aug;10(8):836-41. doi: 10.1111/j.1553-2712.2003.tb00625.x. PMID 12896883
- [Background] Gokel Y, Paydas S, Koseoglu Z, Alparslan N, Seydaoglu G. Comparison of blood gas and acid-base measurements in arterial and venous blood samples in patients with uremic acidosis and diabetic ketoacidosis in the emergency room. Am J Nephrol. 2000 Jul-Aug;20(4):319-23. doi: 10.1159/000013607. PMID 10970986
- [Background] Middleton P, Kelly AM, Brown J, Robertson M. Agreement between arterial and central venous values for pH, bicarbonate, base excess, and lactate. Emerg Med J. 2006 Aug;23(8):622-4. doi: 10.1136/emj.2006.035915. PMID 16858095
- [Background] Chu YC, Chen CZ, Lee CH, Chen CW, Chang HY, Hsiue TR. Prediction of arterial blood gas values from venous blood gas values in patients with acute respiratory failure receiving mechanical ventilation. J Formos Med Assoc. 2003 Aug;102(8):539-43. PMID 14569318
- [Background] Brandenburg MA, Dire DJ. Comparison of arterial and venous blood gas values in the initial emergency department evaluation of patients with diabetic ketoacidosis. Ann Emerg Med. 1998 Apr;31(4):459-65. doi: 10.1016/s0196-0644(98)70254-9. PMID 9546014
- [Background] Ak A, Ogun CO, Bayir A, Kayis SA, Koylu R. Prediction of arterial blood gas values from venous blood gas values in patients with acute exacerbation of chronic obstructive pulmonary disease. Tohoku J Exp Med. 2006 Dec;210(4):285-90. doi: 10.1620/tjem.210.285. PMID 17146193
- [Background] Malatesha G, Singh NK, Bharija A, Rehani B, Goel A. Comparison of arterial and venous pH, bicarbonate, PCO2 and PO2 in initial emergency department assessment. Emerg Med J. 2007 Aug;24(8):569-71. doi: 10.1136/emj.2007.046979. PMID 17652681